CLINICAL TRIAL: NCT04532125
Title: First-In-Human, Randomized, Double-Blinded, Placebo-Controlled Trial in Healthy Subjects to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single and Multiple Ascending Intravenous and Subcutaneous Doses of ARGX-117 Co-mixed With rHuPH20
Brief Title: SAD and MAD Study With IV and SC Doses of ARGX-117
Acronym: ARGX-117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: ARGX-117-1901
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ARGX-117 IV (Experimental): Subjects receiving ARGX-117 IV
  Interventions: Biological: ARGX-117
- Placebo IV (Placebo Comparator): Subjects receiving placebo IV
  Interventions: Other: Placebo
- ARGX-117 PH20 SC (Experimental): Subjects receiving ARGX-117 PH20 SC
  Interventions: Biological: ARGX-117 PH20 SC
- Placebo PH20 SC (Placebo Comparator): Subjects receiving placebo PH20 SC
  Interventions: Other: Placebo PH20 SC
- ARGX-117 + rHuPH20 (Experimental): Subjects receiving ARGX-117 + rHuPH20
  Interventions: Biological: ARGX-117 + rHuPH20
- Placebo + rHuPH20 (Placebo Comparator): Subjects receiving placebo + rHuPH20
  Interventions: Other: placebo + rHuPH20

INTERVENTIONS:
Biological: ARGX-117 — Subjects treated with ARGX-117
  Arms: ARGX-117 IV
Other: Placebo — Subjects treated with placebo
  Arms: Placebo IV
Biological: ARGX-117 + rHuPH20 — Subjects treated with ARGX-117 + rHuPH20
  Arms: ARGX-117 + rHuPH20
Other: placebo + rHuPH20 — Subjects treated with placebo + rHuPH20
  Arms: Placebo + rHuPH20
Biological: ARGX-117 PH20 SC — Subjects treated with ARGX-117 PH20 SC
  Arms: ARGX-117 PH20 SC
Other: Placebo PH20 SC — Subjects treated with placebo PH20 SC
  Arms: Placebo PH20 SC

SUMMARY:
This is a phase 1, first-in-human, double-blinded, randomized, placebo-controlled, escalating single and multiple dose levels trial to evaluate the safety, pharmacokinetics, pharmacodynamics, and immunogenicity of ARGX-117 administered IV and/or SC. Up to 112 healthy, adult male and female subjects of non-childbearing potential will be enrolled in this trial.

ELIGIBILITY:
Inclusion criteria:

1. The subject is between 18 to 65 years of age, inclusive, at the time the informed consent form (ICF) is signed.
2. The subject is either male, or female of nonchildbearing potential. Females in the following categories are considered a woman of nonchildbearing potential:

   1. Postmenopausal female: A postmenopausal state is defined as continuous amenorrhea for at least 1 year without an alternative medical cause and a follicle-stimulating hormone (FSH) measurement of >40 IU/L. A historical pretreatment FSH measurement of>40 IU/L is accepted as proof of a postmenopausal state for subjects on hormone replacement therapy.
   2. Surgically sterile female: women who have had a documented permanent sterilization procedure (ie, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).
3. Female subjects must have a negative serum pregnancy test on day -1 before IMP can be administered.
4. The subject has a body mass index (BMI) within the range 18 to 30 kg/m2 and body weight 50 to 100 kg (inclusive) before IMP administration.
5. The subject is able to understand the requirements of the study and provide written informed consent (including consent for the use and disclosure of research-related health information), and is willing and able to comply with the study protocol procedures (including the required study visits).
6. The subject is in good physical and mental health, per the opinion of the investigator, based on medical history; physical examination findings; ECG recordings; vital sign measurements; systemic lupus erythematous (SLE) panel results; and biochemistry, hematology, INR, and urinalysis laboratory test results prior to the first dose of IMP on day 1.
7. Nonsterilized male subjects who are sexually active with a female partner of childbearing potential must use effective contraception from the signing of the ICF through 260 days after the last IMP administration. A male subject practicing true sexual abstinence (as consistent with the preferred and usual lifestyle) can be included. Sterilized male subjects who have had a vasectomy and with documented absence of sperm post-procedure can be included. Male subjects are not allowed to donate sperm from signing of the ICF through 260 days after the last dose of IMP.
8. The subject has abdominal skin that, in the opinion of the investigator, allows for the absorption and localized safety assessment of SC administration (applicable for dose levels with SC administration only).
9. The subject agrees to discontinue and refrain from the use of all medications, including nonprescription and/or prescription medications, for at least 2 weeks before the first dose of IMP through the EOS visit on day 260 (Part A [SAD]), day 288 (Part B [MAD], cohorts 1 through 5). The occasional use of paracetamol at doses up to 2 g/day with a maximum of 10 g/2 weeks is allowed upon approval from the investigator. COVID-19 immunization recommendations are described in Section 4.3.1.1.
10. The subject is a nonsmoker and does not use any nicotine-containing products. A nonsmoker is defined as an individual who has abstained from smoking for at least 3 months prior to screening.
11. The subject has a negative urine drug and alcohol screen for amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, tricyclic antidepressants and alcohol at screening and on day -1.
12. The subject has a body temperature of 35.5 °C to 37.6 °C at screening and prior to the first dose of IMP day 1.

Exclusion criteria:

1. The subject has a known hypersensitivity to any of the components of the IMP, or, in the opinion of the investigator, a history of a significant allergic reaction to any drug.
2. The subject has previously participated in a clinical study with efgartigimod and was administered an IMP.
3. The subject has a positive serum test at screening for an active viral infection with any of the following conditions:

   1. Hepatitis B virus (HBV) that is indicative of an acute or chronic infection (https://www.cdc.gov/hepatitis/HBV/PDFs/SerologicChartv8.pdf)
   2. Hepatitis C virus (HCV) based on HCV antibody assay
   3. Human immunodeficiency virus
4. The subject tests positively at screening for SLE as determined by the SLE test panel.
5. The subject has a known family history of SLE.
6. The subject has known clinically relevant immunological disorders.
7. The subject has a history of severe allergic or anaphylactic reactions.
8. The subject has clinical evidence of significant serious diseases, underwent a recent major surgery, or has any other condition that, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk. The conditions and diseases that will lead to subject exclusion include recognized uncontrolled risk factors associated with acute respiratory distress syndrome (ARDS) and death in subjects with COVID-19 (eg, hypertension, diabetes, asthma, or chronic obstructive pulmonary disease [COPD]).
9. The subject has a clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection at screening.
10. The subject has the presence or sequelae of gastrointestinal, liver, kidney, or other conditions known to potentially interfere with the absorption, distribution, metabolism, or excretion of IMP.
11. The subject has an estimated glomerular filtration rate of <80 mL/min/1.73 m² (calculated per the Chronic Kidney Disease Epidemiology Collaboration method) at screening.
12. The subject has a history of malignancy except for:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
13. The subject has known genetic deficiencies for the complement cascade system.
14. The subject has clinically relevant abnormalities detected on an ECG that are related to either rhythm or conduction (eg, QTcF >450 ms for male and QTcF >470 ms for female subjects, or a known long QT syndrome).
15. The subject has clinically relevant vital sign abnormalities before the first dose of IMP.
16. The subject had significant blood loss, including blood donation >500 mL, or transfusion of any blood product within 12 weeks before the first dose of IMP, or the subject has a scheduled transfusion within 4 weeks after the end of the study.
17. The subject has received treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months before the first dose of IMP.
18. The subject has a history of any of the following:

    1. consuming more than 21 units of alcoholic beverages per week (Note: 1 unit is 330 mL of beer, 110 mL of wine, or 28 mL of spirits)
    2. alcoholism or drug, chemical, substance abuse within 2 years before screening
    3. consuming a large quantity (>6 cups per day) of coffee, tea, or the equivalent in the 4 weeks before the first dose of IMP.
19. The subject is concurrently participating or has participated, within 90 days before the first dose of IMP or, if known, 5 half-lives of the investigational drug (whichever is longer), in any drug/device or biologic investigational research study.
20. The subject has been administered any systemic immunosuppressant agent within 6 months prior to the first dose of IMP.
21. The subject has been administered any systemic steroid within 3 months prior to the first dose of IMP.
22. The subject is an investigator, subinvestigator, research assistant, pharmacist, study coordinator, or other staff or relative of study personnel directly involved with the conduct of the study.
23. The subject has any condition or circumstances that, in the opinion of the investigator, may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.
24. The subject is a pregnant or lactating female, or intends to become pregnant during the study or within 260 days after the last dose of IMP.
25. The subject has any condition that impairs phlebotomy.
26. The subject has a positive nasopharyngeal polymerase chain reaction (PCR) test for SARS-CoV-2 on day -2 or -1.
27. The subject has any contact with anyone who has tested positive for SARS-CoV-2 or COVID-19 within the last 2 weeks prior to admission to the clinical research center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Number of (S)AE | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)

SECONDARY OUTCOMES:
Area Under The Curve (AUC) | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)
Maximum serum concentrations (Cmax) | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)
  Maximum observed serum concentration
Time to reach maximum serum concentrations (Tmax) | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)
  Time calculated to reach Cmax
Free C2 concentration | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)
  Functional complement activity
Total C2 concentration | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)
  Functional complement activity
CH50 titers | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)
  Functional complement activity
Level of anti-drug antibodies | Up to 37 weeks (arm 1) and up to 42 weeks (arm 2)
  Immunogenicity against ARGX-117

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Site 1, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided